CLINICAL TRIAL: NCT01652924
Title: Efficacy and Safety of Pressure-controlled Ventilation Compared With Manual Ventilation to Reduce Gastric Insufflation During Induction of Anesthesia in Children: Controlled Trial Randomized, Double-blind
Brief Title: Efficacy of Mechanical Ventilation With Facial Mask to Reduce Gastric Insufflation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Olga Luci-a Giraldo Salazar, MD, Anesthesiologist, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Anestesia002
Record Dates: First submitted 2012-07-24; First posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Gastric Insufflation
Keywords: mechanical ventilation; manual ventilation
MeSH Terms: interventions — Respiration, Artificial

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mechanical ventilation (Experimental): 1: Active Comparator Children 1 month-14 years of age Intervention:Mechanical ventilation with facial mask during anesthetic induction
  Interventions: Device: Mechanical ventilation with facial mask
- Manual ventilation (Active Comparator): 2: Active Comparator Children 1 month-14 years of age Intervention: Manual ventilation with facial mask during anesthetic induction
  Interventions: Device: Manual ventilation with facial mask

INTERVENTIONS:
Device: Mechanical ventilation with facial mask — This group includes patients with the randomization process are assigned to mechanical ventilation with facial mask during induction of anesthesia, which will be maintained until to secure airway with endotracheal tube to determine the presence of gastric insufflation. The size of the facial mask is used according to the age and ventilation parameters are: inspiratory pressure 10 cmH2O, PEEP 5 cmH2O, respiratory frequency and relation I/E according to age .
  Other Names: Mechanical ventilation during anesthetic induction
  Arms: Mechanical ventilation
Device: Manual ventilation with facial mask — This group includes patients with the randomization process are allocated to manual ventilation with facial mask during induction of anesthesia, which will be maintained until to secure airway with endotracheal tube to determine the presence of gastric insufflation.
  The size of the facial mask is used according to the age and ventilator y parameters are selected by the anesthesiologist.
  Other Names: Manual ventilation during anesthetic induction
  Arms: Manual ventilation

SUMMARY:
The purpose of this study is to determine whether mechanical ventilation with facial mask during induction anesthesia in the population of 1month to 14years is associated with less risk of gastric insufflations as compared with manual ventilation.

DETAILED DESCRIPTION:
Manual ventilation is the most widely used during induction of anesthesia because of unsupported theoretical advantages in clinical trials as a test of airway patency and adequate ventilation and lung expansion. Additionally, in developing countries until recently lacked sufficient ventilation from supplying controlled fans with different modes that could be used during induction of anesthesia. However, case reports in pediatric and adult patients not intubated, note that manual ventilation could be related to increased frequency of gastric insufflation and predispose to regurgitation and aspiration, impaired ventilation, respiratory failure, reduced cardiac output and rupture or visceral ischemia. To date, no controlled clinical trials have to corroborate or not these experiences.

Gastric insufflation may appear as a result of manual ventilation or mechanical. In connection with the first because it does not allow volume control currents, the time of insufflation or inspiratory pressures, which determine the maximum peak inspiratory pressure, which is directly proportional to the incidence of this complication. Meanwhile, mechanical ventilation is associated with gastric insufflation when pressures exceed certain limits peak airway. vonGoedecke et al, in a clinical trial of mechanical ventilation (pressure control) against the manual in healthy adults during induction of anesthesia and whose outcome was ventilatory variables, they found that mechanical ventilation was associated with lower peak inspiratory pressures lower airway and peak inspiratory flow rates and tidal volumes and minute lower. They recommend mechanical ventilation during induction of anesthesia as the safe technique.

To make ventilation safer in an unprotected airway, can be considered two strategies: limiting the tidal volume or peak inspiratory pressure limit. Seet and colleagues compared in healthy adults two mechanical ventilation strategies in addition to the manual technique during induction considering a composite endpoint of ventilatory variables and gastric insufflation in a clinical trial. They found that pressure-controlled ventilation was associated with lower peak inspiratory pressure and gastric insufflation less than the other two methods, which suggest that this technique is safer and should be the method of choice for ventilation during apnea patients induction.

Several studies have shown the clinical significance of gastric insufflation during induction of anesthesia in 2009, Paal and colleagues presented the results of two studies in animals: one with them in cardiac arrest and another spontaneous circulation, in the first there was a abdominal compartment syndrome leading to hemodynamic compromise, respiratory, metabolic, and finally multi-organ, in animals with spontaneous circulation, the effects were even worse because there was a reduction in survival and in some gastric insufflation was considered as the cause of heart failure . The authors conclude that gastric insufflation alone can cause heart failure and multiple organ failure occurs much faster the more critical is the patient. , In addition to substantial mechanical cardiopulmonary effects, insufflation of the stomach is a complex problem that can cause regurgitation, aspiration, pneumonia and death. Increases abdominal pressure, elevates the diaphragm, restricts lung movement and thus reduce the compliance of the respiratory system. A reduction in respiratory system compliance may direct further ventilation volume into the stomach when the airway is not protected, thus inducing a vicious circle with each breath, increasing the insufflation of the stomach and decreasing lung ventilation. Added to this the fact that the anesthetic drugs reduce the lower esophageal sphincter pressure and more than 90% of cases in children suction produced in the induction of anesthesia, needless to emphasize the importance of controlling this adverse effect. Control of gastric insufflation by the above would be particularly useful in patients with comorbidities that predispose to regurgitation or cardiac arrest patients.

Children are at greater risk of gastric insufflation during induction of anesthesia because of anatomical and physiological characteristics inherent in the conduct of the respiratory system that promote airway obstruction and the passage of air into the stomach: proportional size of the head and tongue, short neck, small chin, among others. This is compounded by the use of a ventilation without control of parameters such tidal volume, inspiratory time and peak inspiratory pressure, as well as reduction of the lower esophageal sphincter pressure caused by anesthetics and airway devices. It is likely that this increased risk of gastric insufflation is the explanation for the increased incidence of aspiration and respiratory complications found in some studies, particularly during anesthetic induction.

The work of von GoedeckeSeet and are pioneers in this new form of induction of anesthesia with ventilation for the patient safer and more comfortable for the anesthesiologist, using more developed fans that bring new anesthesia machines and allow to get the most out of ventilatory modes that are built. However, lacking adequate methodological designs jobs to validate these techniques in different populations, and one of them is the pediatric population, the characteristics mentioned above would suggest that one of the most favored by this method. Therefore, this paper seeks to establish whether the pressure-controlled ventilation during induction of anesthesia reduces the incidence of gastric insufflation compared with manual ventilation of children aged 1 month to 14 years.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and III children, 1 month-14 years of age
* Children scheduled for surgery or therapeutic procedures under general anesthesia and fasting as defined in the fasting guidelines.
* Responsible adult patients whose accept and sign the informed consent of study.

Exclusion Criteria:

* Patients with limited mouth opening or cervical spine extension and classified as difficult airway
* Respiratory diseases
* Children with orogastric or nasogastric tubes
* Children with gastrostomies
* Patients with pulmonary aspiration risk: morbid obesity, intestinal obstruction, gastrointestinal bleeding, gastroparesis, gastroesophageal reflux.

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Gastric insufflation determined by continuous epigastric auscultation until to secure the airway. | From anesthetic induction until to secure airway with endotracheal tube, an expected average of 5 minutes
  Intervention end up once the anesthesiologist to secure airway patient and during this time the investigator will auscultate the epigastrium

SECONDARY OUTCOMES:
Gastric insufflation determined by aspiration with orogastric tube after to secure the airway | First 3 minutes after to secure airway with endotracheal tube
  Intervention end up once the anesthesiologist to secure airway patient and complete aspiration with orogastric tube.

OTHER OUTCOMES:
Gastric insufflation determined by measurement abdominal circumference until to secure the airway and remove orogastric tube. | Before anesthetic induction until to secure airway with endotracheal tube and to remove orogastric tube, an expected average of 20 minutes
  Intervention end up once the anesthesiologist to secure airway patient and remove orogastric tube.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Lucia Giraldo, MD, Principal Investigator — Antioquia University
Locations (1):
- San Vincent Foundation, San Vincent Hospital, Medellín, Antioquia, Colombia